CLINICAL TRIAL: NCT06826755
Title: Melatonin Effects on Cardiovascular Disease Mechanisms in Midlife Women: A Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Naima Covassin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 24-008966
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: Perimenopause; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): placebo will be taken orally once daily, one hour before bedtime. Placebo will be prepared as capsules of identical appearance and taste, using lactose powder as filler.
  Interventions: Dietary Supplement: Placebo
- Melatonin (Other): Melatonin will be taken orally once daily, one hour before bedtime. The use of melatonin is not experimental but rather to observe its effects vs. placebo on cardiovascular risk measures in perimenopausal women.
  Interventions: Dietary Supplement: Terry Naturally® melatonin 5mg SR

INTERVENTIONS:
Dietary Supplement: Terry Naturally® melatonin 5mg SR — Participants will take SR melatonin 5mg (or placebo) orally 1 hour before bed, for approximately 12 weeks. The study is comparing the effects of melatonin supplementation vs. placebo on cardiovascular risk measures in perimenopausal women.
  Arms: Melatonin
Dietary Supplement: Placebo — Participants will take SR melatonin 5mg (or placebo) orally 1 hour before bed, for approximately 12 weeks. The study is comparing the effects of melatonin supplementation vs. placebo on cardiovascular risk measures in perimenopausal women.
  Arms: Placebo

SUMMARY:
The purpose of this research is to study the effects of 12 weeks of melatonin supplementation compared to placebo in women who are in the menopause transition (perimenopause) and have high blood pressure.

ELIGIBILITY:
Inclusion Criteria

* Age 40-55 years old
* Female individuals with intact uterus and at least one ovary
* Hypertension

  o Defined as a prior diagnosis of hypertension, use of antihypertensive agents, or office SBP/DBP ≥130/80 mmHg
* On stable medical regimen (≥ 2 months) if taking other medications

Exclusion Criteria

* Prescription sleeping medications or melatonin supplementation
* Pregnant or lactating
* Use of tobacco, nicotine or vaping products
* Night shift work
* On prescription aspirin
* Severe lactose intolerance
* History of substance use disorder
* History of suicidal ideation
* History of clinically diagnosed anemia (within the past 5 years) or low hemoglobin levels (<11.6 g/dL) within the past 12 months
* Active cancer
* Severe daytime sleepiness (score >15 at the Epworth Sleepiness Scale [ESS])81
* Current or recent (within the past 2 months) participation in other research studies at the discretion of study investigators
* Inability to provide written consent and/or to speak and read English
* Any other medical, geographic, or social factor making study participation impractical

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Nocturnal Systolic Blood Pressure (SBP) | Measured at baseline and at the end of the 12-week intervention
  Measured using 24-hour ambulatory blood pressure (ABP) monitoring, including nighttime BP levels and nocturnal BP dipping.
Change in Nocturnal Diastolic Blood Pressure (DBP) | Measured at baseline and at the end of the 12-week intervention.
  Measured using 24-hour ambulatory blood pressure (ABP) monitoring, including nighttime BP levels and nocturnal BP dipping.

SECONDARY OUTCOMES:
Change in Oxidative Stress Markers | Measured at baseline and at the end of the 12-week intervention.
  Assessed using Blood and urine samples analyzed by Mayo Clinic Laboratories.

CONTACTS AND LOCATIONS:
Overall Officials: Naima Covassin, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No